CLINICAL TRIAL: NCT02683746
Title: A Repeat-dose Study in Subjects With Type 2 Diabetes Mellitus to Assess the Efficacy, Safety, Tolerability and Pharmacodynamics, of Albiglutide Liquid Drug Product
Brief Title: Safety and Efficacy Study of Albiglutide Liquid Drug Product in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200952
Record Dates: First submitted 2016-01-28; First posted 2016-02-17 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pharmacodynamics; Safety; Albiglutide; Tolerability; Type 2 Diabetes Mellitus; Efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albiglutide active LAI plus Placebo lyophilized DCC PI (Experimental): Subjects will receive 30 milligrams (mg) of albiglutide liquid drug product via auto injector and matching placebo via lyophilized DCC pen injector for 4 weeks. The dose will then be up-titrated to 50mg albiglutide for the remaining 22 weeks of the study. The study treatment will be administered once weekly by subcutaneous injection in the abdomen, thigh, or upper arm.
  Interventions: Drug: Lyophilized albiglutide DCC pen injector matching placebo; Drug: Albiglutide liquid auto-injector
- Albiglutide lyophilized DCC PI plus Placebo LAI (Experimental): Subjects will receive 30mg of albiglutide lyophilized drug product via DCC pen injector and matching placebo via auto injector for 4 weeks. The dose will then be up-titrated to 50mg albiglutide for the remaining 22 weeks of the study. The study treatment will be administered once weekly by subcutaneous injection in the abdomen, thigh, or upper arm.
  Interventions: Drug: Lyophilized albiglutide DCC pen injector; Drug: Albiglutide liquid auto-injector matching placebo

INTERVENTIONS:
Drug: Lyophilized albiglutide DCC pen injector — A fixed-dose, fully disposable pen injector system with a prefilled dual chamber glass cartridge (DCC) containing lyophilized albiglutide (30mg or 50mg) delivering an injection volume of 0.5mL.
  Arms: Albiglutide lyophilized DCC PI plus Placebo LAI
Drug: Lyophilized albiglutide DCC pen injector matching placebo — A fixed-dose, fully disposable pen injector system with a prefilled DCC containing matching placebo delivering an injection volume of 0.5mL
  Arms: Albiglutide active LAI plus Placebo lyophilized DCC PI
Drug: Albiglutide liquid auto-injector — A fixed-dose, single use, disposable auto-injector containing albiglutide liquid (30mg or 50mg) in a prefilled glass syringe. The auto-injector delivers the albiglutide liquid in an injection volume of 0.6 mL for the 30mg dose and 1.0 mL for the 50mg dose.
  Arms: Albiglutide active LAI plus Placebo lyophilized DCC PI
Drug: Albiglutide liquid auto-injector matching placebo — A fixed-dose, single use, disposable auto-injector containing matching placebo in a prefilled glass syringe. The auto-injector delivers the matching placebo in an injection volume of 0.6 mL for the 30mg dose and 1.0 mL for the 50mg dose.
  Arms: Albiglutide lyophilized DCC PI plus Placebo LAI

SUMMARY:
This is a phase III, randomized, double-blind, multicenter, parallel group, repeat-dose, study of 26 weeks duration to evaluate the efficacy, safety, tolerability and pharmacodynamic response of albiglutide liquid drug product relative to the commercial lyophilized drug product. The study will specifically evaluate the potential for immunogenicity (example [e.g.] incidences of anti-drug antibodies [ADA]) and injection site reactions (ISRs).

Albiglutide is a novel analogue of glucagon-like peptide-1 (GLP-1) with a sufficiently long half-life to permit once a week injection. Currently, lyophilized albiglutide and the diluent are provided in a dual chamber cartridge (DCC), single-dose pen injector, requiring reconstitution prior to use. A liquid formulation of albiglutide will enable the commercialization of a liquid product in a single dose, ready-to-use prefilled syringe in an auto-injector.

The primary hypothesis of this study is to test that liquid drug product will provide glycemic control (as measured by HbA1c change from baseline) non-inferior to lyophilized drug product for a period of 26 weeks of treatment in subjects with T2DM.

This study will comprise of 3 study periods : screening (2 weeks), treatment (26 weeks) and for those subjects not entering the extension study a follow-up period (8 weeks). Approximately 300 subjects will be randomized in a 1:1 ratio to either Albiglutide active liquid auto-injector (LAI) plus Placebo lyophilized DCC pen injector (lyophilized DCC PI); or, Albiglutide lyophilized DCC PI plus Placebo LAI.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age inclusive
* Historical diagnosis of type 2 diabetes mellitus (T2DM) (at least 3 months), experiencing inadequate glycemic control on current regimen of diet and exercise or on a stable maximal tolerated dose of metformin, maintained for approximately 8 weeks prior to screening.
* HbA1c >=7.0 percent (%) and <=10%.
* Hemoglobin >=11 grams per deciliter (g/dL) (>=110 grams per liter [g/L]) for males and >=10 g/dL (>=100 g/L) for females.
* Body mass index <=40 kilograms per squared meter (kg/m^2)
* Male or female
* Able and willing to provide informed consent.

Exclusion Criteria:

* Type 1 diabetes mellitus
* History of cancer that has not been in full remission for at least 3 years before screening. (A history of squamous cell or basal cell carcinoma of the skin or treated cervical intra-epithelial neoplasia I or II is allowed).
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2.
* History of acute or chronic pancreatitis.
* History of thyroid dysfunction or an abnormal (i.e., outside the normal reference range) thyroid function test assessed by thyroid stimulating hormone at screening.
* Severe gastroparesis, i.e., requiring regular therapy within 6 months before screening.
* History of significant gastrointestinal (GI) surgery that in the opinion of the investigator is likely to significantly affect upper GI or pancreatic function
* History of severe hypoglycemia unawareness
* Diabetic complications or any other clinically significant abnormality .
* Clinically significant Cardiovascular (CV) and/or cerebrovascular disease within 3 months before screening
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 470 milliseconds (msec).
* ALT >2.5x upper limit of the normal range (ULN) or bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* Estimated glomerular filtration rate (eGFR) <=30 milliliter (mL)/minute (min)/1.73 squared meter (m^2) (calculated using the Modification of Diet in Renal Disease [MDRD] formula) at screening.
* Fasting triglyceride level >750 milligrams per deciliter (mg/dL) at screening.
* Hemoglobinopathy that may affect proper interpretation of HbA1c.
* Medical or psychiatric disorders that would preclude effective participation in study.
* Use of oral or systemically injected glucocorticoids within the 3 months before randomization or high likelihood of a requirement for prolonged treatment (>1 week) in the 6 months following randomization.
* Use of dipeptidyl peptidase-IV inhibitors within the 3 months before randomization.
* History of alcohol or substance abuse within one year before screening.
* Known allergy to albiglutide or any product components (including yeast and human albumin), any other glucagon-like peptide-1 (GLP-1) analogue, or other study medication's excipients OR other contraindications (per the prescribing information) for the use of potential study medications.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (65):
- United States (65):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Canyon Country, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Lomita, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Van Nuys, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Brooksville, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fleming Island, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Conyers, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Elgin, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Norwood, Ohio
  - GSK Investigational Site, Perrysburg, Ohio
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Pharr, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Spring, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Federal Way, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=200952

REFERENCES:
- [Background] Shaddinger BC, Soffer J, Vlasakakis G, Shabbout M, Weston C, Nino A. Efficacy and safety of an albiglutide liquid formulation compared with the lyophilized formulation: A 26-week randomized, double-blind, repeat-dose study in patients with type 2 diabetes mellitus. Diabetes Res Clin Pract. 2019 Jun;152:125-134. doi: 10.1016/j.diabres.2019.04.018. Epub 2019 Apr 18. PMID 31004676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This repeat-dose study of albiglutide was conducted at 153 sites in the United States (US). A total of 624 participants with type 2 diabetes mellitus (T2DM) were screened; of these 316 were screen failures and 308 were randomized to receive albiglutide liquid drug product or lyophilized drug product in a 1:1 ratio.
Groups:
- Albiglutide Liquid: Eligible participants received 30 milligrams (mg) of albiglutide active liquid auto-injector along with placebo lyophilized dual chamber cartridge (DCC) pen injector once weekly for 4 weeks by subcutaneous (SC) injection in the abdomen, thigh, or upper arm. After 4 weeks, albiglutide dose was up-titrated to 50 mg for the remaining 22 weeks of the study treatment period.
- Albiglutide Lyophilized: Eligible participants received 30 mg of albiglutide active lyophilized DCC pen injector along with placebo liquid auto-injector once weekly for 4 weeks by SC injection in the abdomen, thigh, or upper arm. After 4 weeks, albiglutide dose was up-titrated to 50 mg for the remaining 22 weeks of the study treatment period.
Period: Overall Study
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Started | 154 | 154
Completed | 138 | 140
Not Completed | 16 | 14
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: One participant was randomized to receive Albiglutide and withdrawn from the study prior to receiving any study medication for reason 'withdrew consent'.
Groups:
- Total: Total of all reporting groups
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized | Total
Number analyzed (Participants) | 153 | 154 | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (9.25) | 56.6 (10.08) | 57.1 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 79 | 149
  Male | 83 | 75 | 158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity customized: American Indian (AI) or Alaska native Heritage | 1 | 3 | 4
  Race/ethnicity customized: Asian- Central/ South Asian Heritage | 1 | 0 | 1
  Race/ethnicity customized: Asian- Japanese/East Asian (EA)/South EA Heritage | 2 | 2 | 4
  Race/ethnicity customized: Black or African American (AA) Heritage | 15 | 24 | 39
  Race/ethnicity customized: Native Hawaiian or Other Pacific Islander Heritage | 1 | 1 | 2
  Race/ethnicity customized: White Heritage | 129 | 122 | 251
  Race/ethnicity customized: Multiple- AI or Alaska Native and White Heritage | 2 | 1 | 3
  Race/ethnicity customized: Multiple- Black or AA and White Heritage | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 26
Description: Blood samples will be collected from participants at specific time points to evaluate HbA1c to monitor for potential hyperglycemia. The last measurement collected prior to the first dose of randomized study treatment was considered as Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was performed using a mixed-effect model with repeated measures (MMRM) method. The primary analysis will include all HbA1c values collected at scheduled visits from Week 4 up to Week 26. This will include values after hyperglycemia rescue and discontinuation from investigational product. Imputation under the non-inferiority null hypothesis for missing data will be incorporated.
Time Frame: Baseline and Week 26
Population: Intent-To-Treat (ITT) Population comprised of all randomized participants who received at least one dose of study treatment and have a Baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: Percentage of total hemoglobin
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 153 | 154
Percentage of total hemoglobin | -1.12 (0.072) | -1.18 (0.072)
Statistical Analysis 1: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Non-Inferiority — The primary hypothesis tested was that the liquid drug product would provide glycemic control non-inferior to the lyophilized drug product for a period of 26 weeks of treatment in participants with T2DM. Non-inferiority testing was performed at a one-sided alpha of 0.025 and non-inferiority margin of 0.4; p = 0.0002, MMRM model — P-value from a one-sided t-test to test whether the difference of least square means (Albiglutide liquid - Albiglutide lyophilized) is equal to the pre-specified non-inferiority margin of 0.4%; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.13 to 0.24]

2. Secondary Outcome: Number of Participants With On-therapy Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect, other situations and is associated with liver injury or impaired liver function.
Time Frame: Up to Week 26
Population: Safety Population comprised of all enrolled participants who received at least one dose of study treatment.
Measure: Number; unit: Participnats
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 153 | 154
Participnats
  AEs | 101 | 94
  SAEs | 7 | 9

3. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters of Potential Clinical Concern (PCC)
Description: Chemistry parameters for which PCC values were identified were alanine aminotransferase (ALT) (if value >3 * upper limit of normal [ULN]), albumin (if value >5 gram/liter [g/L] above ULN or below lower limit of normal [LLN]), alkaline phosphatase (alk.phosph.) (if value >3*ULN), aspartate aminotransferase (AST) (if value >3*ULN), total bilirubin (if value >1.5 ULN), calcium (if value <1.8 or >3.0 millimoles per liter [mmol/L]), carbon di oxide (CO2) (if value <16 or >40 mmol/L), creatinine (if value >159 micromoles per liter [µmol/L]), direct bilirubin (if value >1.35*ULN), gamma glutamyl transferase (GGT) (if value >3*ULN), potassium (if value >0.5 mmol/L below LLN and >1.0 mmol/L above ULN), protein (if value >15 g/L above ULN or below LLN), sodium (>5 mmol/L below LLN or above ULN), urate (if value >654 µmol/L) and urea (if value >2*ULN). Number of participants with chemistry parameters of PCC at 'any visit post-Baseline' are presented.
Time Frame: Up to Week 26
Population: Safety Population. Only those participants present at 'any visit post-Baseline' are analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 153 | 153
Participants
  ALT; >3*ULN | 0 | 1
  Albumin; >5 g/L below LLN | 0 | 0
  Albumin; >5 g/L above ULN | 0 | 0
  Alk.phosph.; >3*ULN | 0 | 0
  AST; >3*ULN | 1 | 1
  Bilirubin; >1.5*ULN | 0 | 2
  Calcium; <1.8 mmol/L | 0 | 0
  Calcium; >3.0 mmol/L | 1 | 0
  CO2; <16 mmol/L | 1 | 6
  CO2; >40 mmol/L | 0 | 0
  Creatinine; >159 µmol/L | 1 | 1
  Direct bilirubin; >1.35ULN | 0 | 1
  GGT; >3*ULN | 1 | 4
  Potassium; >0.5 mmol/L below LLN | 0 | 1
  Potassium; >1.0 mmol/L above ULN | 0 | 1
  Protein; >15 g/L below LLN | 0 | 0
  Protein; >15 g/L above ULN | 0 | 0
  Sodium; >5 mmol/L below LLN | 1 | 0
  Sodium; >5 mmol/L above ULN | 0 | 2
  Urate; >654 µmol/L | 1 | 1
  Urea; >2*ULN | 0 | 0

4. Secondary Outcome: Number of Participants With Hematology Parameters of PCC
Description: Hematology parameters for which PCC values were identified were hematocrit (if value >0.05 below LLN or >0.04 above ULN), Hemoglobin (Hb) (if value >20 g/L below LLN or >10 g/L above ULN), lymphocytes (if value <0.5*LLN), neutrophils (if value <1 giga unit per liter [GI/L]) and platelets (if value <80 GI/L or >500 GI/L). Number of participants with hematology parameters of PCC at 'any visit post-Baseline' are presented.
Time Frame: Up to Week 26
Population: Safety Population. Only those participants present at 'any visit post-Baseline' are analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 153 | 153
Participants
  Hematocrit; >0.05 (fraction of 1) below LLN | 2 | 6
  Hematocrit; >0.04 (fraction of 1) above ULN | 5 | 2
  Hb; >20 g/L below LLN | 3 | 9
  Hb; >10 g/L above ULN | 2 | 2
  Lymphocytes; <0.5*LLN | 0 | 0
  Neutrophils; <1 GI/L | 1 | 0
  Platelets; <80 GI/L | 0 | 0
  Platelets; >500 GI/L | 1 | 1

5. Secondary Outcome: Number of Participants With Vital Signs of PCC
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate were measured in a seated position after at least 5 minutes of rest. SBP values <100 millimeters of mercury (mmHg) and >170 mmHg, DBP values <50 mmHg and >110 mmHg, pulse rate values <50 beats per minute (bpm) and >120 bpm were considered as PCC values. Number of participants with PCC values of vital signs for 'any visit post-Baseline' are presented.
Time Frame: Up to Week 34
Population: Safety Population. Only those participants present at 'any visit post-Baseline' are analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 153 | 153
Participants
  SBP: <100 mmHg | 18 | 16
  SBP; >170 mmHg | 11 | 13
  DBP; <50 mmHg | 0 | 0
  DBP; > 110 mmHg | 3 | 3
  Pulse rate; < 50 bpm | 5 | 2
  Pulse rate; > 120 bpm | 1 | 0

6. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Parameters of PCC
Description: Single measurements of 12-lead ECG were obtained in semi recumbent position using an ECG machine that automatically calculates the heart rate and measures PR and QT interval corrected for heart rate according to Fridericia's formula (QTcF). Number of participants with ECG values of PCC at 'any visit post-Baseline' are presented. ECG mean heart rate values <50 or >120, PR interval >300 milliseconds (msec), QRS interval >200 msec, QTcF interval >=500 msec were considered as PCC values. Number of participants with PCC values of ECG parameters for 'any visit post-Baseline' are presented.
Time Frame: Up to Week 26
Population: Safety Population. Only those participants present at 'any visit post-Baseline' are analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 152 | 152
Participants
  ECG mean heart rate; <50 bpm | 2 | 2
  ECG mean heart rate; >120 bpm | 1 | 0
  PR interval; >300 msec | 1 | 2
  QRS duration; >200 msec | 0 | 0
  QTcF interval; >=500 msec | 0 | 0

7. Secondary Outcome: Number of Participants With Positive Result for Anti-albiglutide Antibody
Description: Blood samples were obtained from participants at specific time points before administration of study treatment. The presence of anti-albiglutide antibodies was assessed using a validated enzyme linked immunosorbent assay (ELISA). The assay involves screening, confirmation, and titration steps (tiered-testing approach). Number of participants with positive anti- albiglutide antibody results at 'any visit post-Baseline' are presented.
Time Frame: Up to Week 34
Population: Safety Population. Only those participants present at 'any visit post-Baseline' are analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 152 | 152
Participants | 17 | 16

8. Secondary Outcome: Number of Participants With Injection Site Reactions (ISR)
Description: Number of participants with ISR incidences were evaluated at specific time points. Each week included those participants with the onset of an ISR during that particular week as well as those participants with ISR from previous weeks that have not resolved.
Time Frame: Up to Week 34
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 153 | 154
Participants | 17 | 18

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: Blood samples were collected from participants at specific time points to evaluate FPG to monitor for potential hyperglycemia. The last measurement collected prior to the first dose of randomized study treatment was considered as Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was performed using a MMRM model.
Time Frame: Baseline and Week 26
Population: ITT Population. Only those participants available at Week 26 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Mmol/L
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 141 | 136
Mmol/L | -2.22 (0.191) | -1.88 (0.195)
Statistical Analysis 1: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.83 to 0.14]

10. Secondary Outcome: Change From Baseline in HbA1c Over Time
Description: Blood samples were collected from participants at specific time points to evaluate HbA1c to monitor for potential hyperglycemia. The last measurement collected prior to the first dose of randomized study treatment was considered as Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was performed using a MMRM model and model-adjusted least square mean (LS mean) and standard error have been presented. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 26
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent of total hemoglobin
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 153 | 154
Percent of total hemoglobin
  Week 4; n= 148, 149: number analyzed (Participants) | 148 | 149
  Week 4; n= 148, 149 | -0.50 (0.045) | -0.54 (0.046)
  Week 8; 145, 147: number analyzed (Participants) | 145 | 147
  Week 8; 145, 147 | -0.96 (0.057) | -1.02 (0.057)
  Week 12; n= 137, 145: number analyzed (Participants) | 137 | 145
  Week 12; n= 137, 145 | -1.15 (0.065) | -1.23 (0.064)
  Week 16; n= 136, 144: number analyzed (Participants) | 136 | 144
  Week 16; n= 136, 144 | -1.25 (0.070) | -1.27 (0.070)
  Week 20; n= 137, 142: number analyzed (Participants) | 137 | 142
  Week 20; n= 137, 142 | -1.24 (0.067) | -1.26 (0.066)
  Week 26; n= 138, 141: number analyzed (Participants) | 138 | 141
  Week 26; n= 138, 141 | -1.16 (0.071) | -1.17 (0.071)
Statistical Analysis 1: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; p < 0.0001, MMRM model — Calculated P-value from a one-sided t-test to test whether the difference of least square means (Albiglutide liquid - Albiglutide lyophilized) is equal to the pre-specified non-inferiority margin of 0.4%; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.07 to 0.13] — Difference in HbA1c levels between albiglutide liquid and lyophilized product at Week 4 are presented
Statistical Analysis 2: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; p < 0.0001, MMRM model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.07 to 0.20] — Difference in HbA1c levels between albiglutide liquid and lyophilized product at Week 8 are presented
Statistical Analysis 3: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; p < 0.0001, MMRM model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.08 to 0.24] — Difference in HbA1c levels between albiglutide liquid and lyophilized product at Week 12 are presented
Statistical Analysis 4: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; p < 0.0001, MMRM model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.16 to 0.20] — Difference in HbA1c levels between albiglutide liquid and lyophilized product at Week 16 are presented
Statistical Analysis 5: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; p < 0.0001, MMRM model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.15 to 0.19] — Difference in HbA1c levels between albiglutide liquid and lyophilized product at Week 20 are presented
Statistical Analysis 6: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; p < 0.0001, MMRM model — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.17 to 0.20] — Difference in HbA1c levels between albiglutide liquid and lyophilized product at Week 26 are presented

11. Secondary Outcome: Change From Baseline in FPG Over Time
Description: Blood samples were collected from participants at specific time points to evaluate FPG to monitor for potential hyperglycemia. The last measurement collected prior to the first dose of randomized study treatment was considered as Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was performed using a MMRM model. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 26
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Mmol/L
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 153 | 154
Mmol/L
  Week 1; n= 148, 144: number analyzed (Participants) | 148 | 144
  Week 1; n= 148, 144 | -1.04 (0.165) | -1.29 (0.167)
  Week 2; n= 143, 145: number analyzed (Participants) | 143 | 145
  Week 2; n= 143, 145 | -1.52 (0.180) | -1.77 (0.181)
  Week 3; n= 145, 140: number analyzed (Participants) | 145 | 140
  Week 3; n= 145, 140 | -1.71 (0.168) | -1.70 (0.170)
  Week 4; n= 142, 145: number analyzed (Participants) | 142 | 145
  Week 4; n= 142, 145 | -1.93 (0.162) | -1.91 (0.164)
  Week 5; n= 146, 143: number analyzed (Participants) | 146 | 143
  Week 5; n= 146, 143 | -2.04 (0.160) | -2.23 (0.162)
  Week 6; n= 145, 145: number analyzed (Participants) | 145 | 145
  Week 6; n= 145, 145 | -2.07 (0.167) | -2.22 (0.169)
  Week 7; n= 146, 144: number analyzed (Participants) | 146 | 144
  Week 7; n= 146, 144 | -1.93 (0.176) | -2.20 (0.179)
  Week 8; n= 143, 141: number analyzed (Participants) | 143 | 141
  Week 8; n= 143, 141 | -2.19 (0.169) | -2.38 (0.171)
  Week 9; n= 142, 141: number analyzed (Participants) | 142 | 141
  Week 9; n= 142, 141 | -2.05 (0.178) | -2.08 (0.180)
  Week 10; n= 141, 142: number analyzed (Participants) | 141 | 142
  Week 10; n= 141, 142 | -2.03 (0.173) | -2.17 (0.175)
  Week 11; n= 141, 139: number analyzed (Participants) | 141 | 139
  Week 11; n= 141, 139 | -2.01 (0.181) | -2.12 (0.184)
  Week 12; n= 137, 137: number analyzed (Participants) | 137 | 137
  Week 12; n= 137, 137 | -2.16 (0.176) | -2.19 (0.178)
  Week 13; n= 140, 136: number analyzed (Participants) | 140 | 136
  Week 13; n= 140, 136 | -2.04 (0.202) | -2.09 (0.205)
  Week 16; n= 140, 140: number analyzed (Participants) | 140 | 140
  Week 16; n= 140, 140 | -2.02 (0.189) | -2.09 (0.191)
  Week 20; n= 139, 134: number analyzed (Participants) | 139 | 134
  Week 20; n= 139, 134 | -1.87 (0.197) | -1.90 (0.201)
  Week 26; n= 141, 136: number analyzed (Participants) | 141 | 136
  Week 26; n= 141, 136 | -2.22 (0.191) | -1.88 (0.195)
Statistical Analysis 1: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.15 to 0.65] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 1 are presented
Statistical Analysis 2: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.20 to 0.69] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 2 are presented
Statistical Analysis 3: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.42 to 0.40] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 3 are presented
Statistical Analysis 4: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.42 to 0.36] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 4 are presented
Statistical Analysis 5: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.19, 95% CI 2-sided [-0.19 to 0.57] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 5 are presented
Statistical Analysis 6: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.26 to 0.55] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 6 are presented
Statistical Analysis 7: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.27, 95% CI 2-sided [-0.16 to 0.71] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 7 are presented
Statistical Analysis 8: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.19, 95% CI 2-sided [-0.22 to 0.60] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 8 are presented
Statistical Analysis 9: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.41 to 0.47] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 9 are presented
Statistical Analysis 10: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.28 to 0.57] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 10 are presented
Statistical Analysis 11: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.34 to 0.56] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 11 are presented
Statistical Analysis 12: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.41 to 0.46] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 12 are presented
Statistical Analysis 13: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.47 to 0.57] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 13 are presented
Statistical Analysis 14: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.41 to 0.54] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 16 are presented
Statistical Analysis 15: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.47 to 0.53] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 20 are presented
Statistical Analysis 16: Comparison: Albiglutide Liquid vs Albiglutide Lyophilized; Test type: Other; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.83 to 0.14] — Difference in FPG levels between albiglutide liquid and lyophilized product at Week 26 are presented

12. Secondary Outcome: Trough Plasma Concentration of Albiglutide Over Time
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of albiglutide. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose at Week 12 and Week 26
Population: PK Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Albiglutide Liquid | Albiglutide Lyophilized
Number analyzed (Participants) | 151 | 149
Nanograms per milliliter (ng/mL)
  Week 12; n= 127, 130: number analyzed (Participants) | 127 | 130
  Week 12; n= 127, 130 | 3996.9 (1613.02) | 3927.1 (1537.45)
  Week 26; n= 127, 127: number analyzed (Participants) | 127 | 127
  Week 26; n= 127, 127 | 4196.6 (1500.57) | 3929.1 (1338.08)

ADVERSE EVENTS:
Time Frame: On-therapy SAEs and non-SAEs are presented from the start of study treatment up to Week 26.
Description: On-therapy SAEs and non-SAEs are reported for the safety Population, comprised of all enrolled participants who received at least one dose of study treatment.
Arm/Group | Albiglutide Active LAI Plus Placebo Lyophilized DCC PI | Albiglutide Lyophilized DCC PI Plus Placebo LAI
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/154
Serious Adverse Events (participants affected / at risk) | 7/153 | 9/154
Other Adverse Events (participants affected / at risk) | 101/153 | 94/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide Active LAI Plus Placebo Lyophilized DCC PI (N=153) | Albiglutide Lyophilized DCC PI Plus Placebo LAI (N=154)
Angina pectoris (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide Active LAI Plus Placebo Lyophilized DCC PI (N=153) | Albiglutide Lyophilized DCC PI Plus Placebo LAI (N=154)
Upper respiratory tract infection (Infections and infestations) | 8 | 20
Viral upper respiratory tract infection (Infections and infestations) | 10 | 10
Bronchitis (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 2 | 5
Gastroenteritis (Infections and infestations) | 3 | 2
Sinusitis (Infections and infestations) | 1 | 4
Viral infection (Infections and infestations) | 4 | 0
Conjunctivitis (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 2 | 1
Otitis externa (Infections and infestations) | 1 | 2
Tooth abscess (Infections and infestations) | 2 | 1
Tooth infection (Infections and infestations) | 2 | 1
Localised infection (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 1
Papilloma viral infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Vaginal abscess (Infections and infestations) | 0 | 1
Viraemia (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 17 | 25
Diarrhoea (Gastrointestinal disorders) | 15 | 11
Constipation (Gastrointestinal disorders) | 13 | 2
Vomiting (Gastrointestinal disorders) | 6 | 6
Toothache (Gastrointestinal disorders) | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 6
Abdominal distension (Gastrointestinal disorders) | 4 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 1 | 2
Dental caries (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Eructation (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon sheath disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Injection site reaction (General disorders) | 6 | 6
Injection site bruising (General disorders) | 3 | 5
Injection site erythema (General disorders) | 1 | 7
Injection site pruritus (General disorders) | 2 | 5
Injection site rash (General disorders) | 3 | 3
Fatigue (General disorders) | 2 | 3
Pyrexia (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Injection site discolouration (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 1 | 0
Injection site induration (General disorders) | 0 | 1
Injection site irritation (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Injection site swelling (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Vaccination site bruising (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1
Vessel puncture site reaction (General disorders) | 0 | 1
Headache (Nervous system disorders) | 12 | 14
Dizziness (Nervous system disorders) | 6 | 6
Neuropathy peripheral (Nervous system disorders) | 3 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Periodic limb movement disorder (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 4
Laceration (Injury, poisoning and procedural complications) | 1 | 3
Limb injury (Injury, poisoning and procedural complications) | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 8 | 7
Hot flush (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1
Binge eating (Psychiatric disorders) | 0 | 1
Borderline personality disorder (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 2 | 5
Food allergy (Immune system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Mitral valve calcification (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Age-related macular degeneration (Eye disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Oligomenorrhoea (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Heart sounds abnormal (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT02683746/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT02683746/SAP_001.pdf